CLINICAL TRIAL: NCT05560737
Title: ODYSSEE-vCHAT Mental Health Study: A Virtual Community Promoting Health Literacy, Self-Care, and Peer Support for Heart Failure and Kidney Disease
Brief Title: ODYSSEE-vCHAT Mental Health Program for Heart Failure and Kidney Disease Patients
Acronym: ODYSSEEvCHAT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other); Mount Sinai Hospital, Canada (Other); The Ottawa Hospital (Other)
Responsible Party: Principal Investigator, Robert Nolan, Senior Scientist, University Health Network, Toronto
Other Study IDs: 20-6005; MS2173076 (Other Grant/Funding Number: Canadian Institutes of Health Research (CIHR)); 3787 (Other: Sunnybrook Hospital Research Ethics Board); 21-0057-E (Other: Mount Sinai Hospital Research Ethics Board); 20220139-01H (Other: The Ottawa Hospital Research Ethics Board)
Record Dates: First submitted 2021-08-26; First posted 2022-09-29 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Chronic Heart Failure; Chronic Kidney Diseases
Keywords: Digital counselling; Social network support; eHealth; Self-care; Mental health; COVID-19; Cognitive behavioural therapy; Motivational interviewing
MeSH Terms: conditions — Renal Insufficiency, Chronic; Psychological Well-Being; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 16 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: ODYSSEE-vCHAT — ODYSSEE-vCHAT consists of:
  * Automated digital counselling resources (educational pages, videos, tools, and trackers)
  * Chatrooms available 24/7
  * Weekly 30-minute presentations and discussions led by a healthcare professional or patient representative
  Each aspect was informed by a rotating schedule of 7 weekly self-care themes. Webcasts were recorded and streamed to our private YouTube channel, and associated hyperlinks were shared on the program. Subjects had the option of submitting photographs depicting heart-healthy lifestyles and activities (with no identifying, sensitive, or personal information) to the Gallery Wall.
  Subjects were invited by email to access the resources available to them. They logged on to the program using password-protected personal accounts. Each participant's total number of logins and login time (with timestamps) were recorded. Assessments occurred online at baseline, months 4 and 8, and study completion (up to 16 months).

SUMMARY:
INTRODUCTION

Psychological distress and reduced quality of life are prevalent in patients with chronic heart failure (CHF) and advanced chronic kidney disease (CKD). In addition, persons with CHF or CKD live with increased risk of primary or secondary complications associated with COVID-19, including mortality. International task force committees report that medical therapy combined with counselling for CHF and CKD self-care optimizes clinical outcomes. Digital health initiatives present an effective solution in light of the recent issue of declining patient attendance in essential outpatient appointments due to the increased risk of COVID-19 exposure.

HYPOTHESES

At study completion (up to 16 months), it is hypothesized that there will be a significant increase from baseline in the proportion of participants with clinically improved or sustained positive mental health. Additionally, greater engagement with the ODYSSEE-vCHAT program is expected to be linked with improved self-reported health- and wellbeing-related outcomes at months 4 and 8 and study completion (up to 16 months).

RECRUITMENT

Patients with CHF or CKD who are at least 18 years old were recruited from the University Health Network (UHN), Sunnybrook Hospital, Mount Sinai Hospital, The Ottawa Hospital, and the community. Accrual of the sample (N = 215) occurred over a 14-month period.

DESIGN

This is a single group, open label, pre-post study with assessments at baseline, months 4 and 8, and study completion (up to 16 months). ODYSSEE-vCHAT contacted subjects each week inviting them to participate or partake in digital counselling resources, chatrooms, and presentations with group discussions. Participation in supplemental mental health programs was monitored by self-report.

ANALYSES

A binomial logistic regression will evaluate if there is a greater proportion of participants with positive mental health at study completion. This analysis will assess if the proportion of participants with positive mental health at study completion (up to 16 months) is independently associated with ODYSSEE-vCHAT engagement (login minutes). General linear models will test secondary outcomes, adjusting for baseline assessments and potential covariates. Significance in all tests will be p < 0.05, 2-sided. Any unplanned analyses will be adjusted for using the Bonferroni procedure.

DETAILED DESCRIPTION:
BACKGROUND

Mental health needs are pronounced for individuals with CHF or advanced CKD. Clinically significant symptoms of depression and anxiety are prevalent in 22% and 33% of outpatients with CHF, respectively, and 26% and 12-52% of outpatients with CKD, respectively. Two psychosocial factors are known to compound the disease burden experienced by persons with these chronic progressive conditions: Diminished social support and isolation. These factors compromise patients' psychological wellbeing and quality of life, while contributing to caregiver burden or stress. Additionally, persons with CHF or CKD experience an increased risk of exposure to COVID-19 and associated mortality. The impact of the pandemic on mental health includes greater symptoms of anxiety, mood disturbance, social isolation due to social distancing, disruption to sleep or eating patterns, impaired concentration due to stress, and use of drugs or alcohol.

A digital program of social network support that is integrated with automated counselling is central to this proposal. This approach has demonstrated a potential to improve psychological wellbeing and quality of life while reducing social isolation, increase patient engagement with digital programs, and sustain preventive self-care for mental health with positive role modelling, information sharing, and structured presentations. Home-based digital health programs are changing practice standards for outpatient medical care. This development is consistent with task force guidelines for infection prevention and control that advocate for the development of virtual outpatient programs. Digital health initiatives are also well-suited to effectively address the recent problem that patients are declining to attend essential outpatient appointments due to fear of COVID-19 exposure.

The present study will generate novel insights on how to optimize the efficacy and usability of a scalable, evidence-based digital program where social network technology and automated counselling are used synergistically to promote mental health for persons at increased risk for COVID-19.

RATIONALE

Meta-analysis indicates a login rate of only 72% and a mean dropout rate of 15% (range = 0 to 62%) in digital health programs, which undermines population reach. The ODYSSEE-vCHAT proposal is consistent with COVID-19 task force recommendations to develop patient-centered, evidence-based digital interventions that can sustain patient engagement and scale to the wider population to optimize quality of life and mental health. A previous trial of automated digital counselling for CHF increased patient engagement over 12 months by 37% relative to a control group receiving enhanced usual care, and participation was independently associated with improved quality of life. ODYSSEE-vCHAT, with its added social network components, is designed to improve upon this outcome.

HYPOTHESES

The primary hypothesis is that, at completion (up to 16 months), there will be an increase from baseline in the proportion of participants with clinically improved or sustained positive mental health, defined as a "minimally important increase" of ≤ 3.8 points or a score of ≤ 65 on the Mental Component Summary (MCS) of the 36-Item Short-Form Survey.

The secondary hypothesis is that engagement with self-care resources [defined by (i) sum login minutes, (ii) sum logins, and (iii) number of login days prior to a lapse of ≥ 1 month] at months 4 and 8 and study completion] will be independently associated with the following outcomes:

* Decreased depression, anxiety, loneliness, and use of alcohol, nicotine, and cannabis
* Increased psychological wellbeing, health-related quality of life, adherence to self-care behaviours (CHF only), engagement in goal-directed activities for living well, health literacy, active involvement in medical care, perceived social support, and physical functioning

Additionally, participant engagement with self-care resources will be independently and positively associated with the proportion of participants demonstrating improved or sustained positive mental health.

POTENTIAL RISKS

Participants may have experienced discomfort with the following:

* Responding to items in the assessments that are considered personal
* Using ODYSSEE-vCHAT because they are not familiar with the software
* Verbally contributing to the discussion segments of the webcasts as their voice would be recorded
* Submitting an audio or video response to the webcasts because they would no longer be an anonymous participant (audio or video comments may also be used for research and educational purposes in the public domain)

SAFETY PARAMETERS

Refusals to respond to any item(s) posed in the questionnaire packages were accommodated.

Video tutorials on how to use ODYSSEE-vCHAT were provided. Assistance over the telephone was offered when required.

During webcasts, visual input from patients remained disabled to protect their identification. If participants preferred to contribute to the discussion without speaking, they were encouraged to use the chat feature on Zoom instead. Comments written in the chat were not included in the recording of the session.

Participants' audio or video comments were censored for inappropriate comments pertaining to violence, sexual content, coarse language, etc. Regarding videos that were selected for presentation to other participants in the trial, or to the public, patients were notified so that they had an opportunity to grant or withhold their permission for this use of their video.

Social network chatrooms were HIPPA compliant and moderated by three levels of content filtering to ensure that posts meet conventional standards of ethical conduct. Level 1 was a search algorithm that is automatically updated with banned word lists. Level 2 was carried by patient volunteers through self-report. Level 3 was performed by research assistants.

Finally, subjects were offered an opportunity to send the research team photographs via email which depict healthy lifestyles. Patients were asked not to include any identifying, sensitive, or personal information in the photographs, which would be shared with other participants to encourage social interaction. Participants were informed that they may contact the research team at any time to have their photo submissions withdrawn.

STATISTICAL PLAN

Primary outcome:

At study completion, the McNemer c2 test will assess if there is a greater proportion of participants with positive mental health at study completion. A binomial logistic regression will evaluate if the proportion of participants with positive mental health at study completion is independently associated with vCHAT engagement. Covariates will include CHF or CKD diagnosis, reported gender, registered COVID-19 diagnosis, age, income, and participation in a supplemental mental health program.

Secondary outcomes:

General linear models will assess if separate outcomes at months 4, 8, and study completion (up to 16 months) demonstrate a significant therapeutic change in:

* Depression
* Anxiety
* Perceived social support
* Loneliness
* Health-related quality of life
* Adherence to self-care (CHF only)
* Engagement in goal-directed activities for living well
* Health literacy
* Active involvement in medical care
* Use of alcohol, cigarettes, and cannabis

Generalized estimating equation models will assess if the proportion of participants with positive MCS status at study completion is independently associated with ODYSSEE-vCHAT engagement for each subcomponent of digital counselling and social network support across assessments. Covariates will include assessment intervals.

Exploratory outcomes:

Separate analyses will be conducted for gender. The association between engagement with self-care resources and overall mental health will also be analyzed.

DEVIATIONS FROM STATISTICAL PLAN

Since the statistical plan involves exploratory analyses, a need to deviate from was not anticipated. Nevertheless, the Statistical Analysis and Methodology Committee were consulted regularly. Any unplanned analyses will be adjusted using the Bonferroni procedure.

SAMPLE SIZE

A recent study reported a significant 12-month improvement on the MCS for telehealth support versus usual care. Within-group change on the MCS for telehealth was 3.81 (standard deviation = 10.7). The sample size required to replicate this outcome for ODYSSEE-vCHAT is 188. With a recruitment period of 8 months, a minimum follow-up of 3 months, and a 14.7% rate of withdrawal or attrition (based on the CHF-CePPORT trial), the final sample size estimate is 240, (α = 0.05, β = 0.80). However, a total sample size of N = 215 was accrued.

SUBJECT COMPLIANCE

Attendance for assessments was facilitated by telephone and email reminders if a participant failed to complete an assessment within 5 to 7 days of receiving the initial invitation.

SUBJECT WITHDRAWAL

Adverse events such as an unforeseen mental health crisis may have affected a patient's ability to participate in this trial. In cases of patient withdrawal, all data up to this point pertaining to the patient will be used for outcome analyses. The Steering Committee would review how and whether the subject should be replaced in the trial. The referring cardiologist or nephrologist would be alerted about the withdrawal.

QUALITY CONTROL AND ASSURANCE

The Data Review or Monitoring Committee ensured that the trial met an appropriate standard for data quality control. The Steering Committee adjudicated primary and secondary outcomes, as well as reviewed and advised the team about the trial's progress, protocol compliance, and any adverse incidents.

CONSENT

Cardiologists or nephrologists and their nursing staff in participating outpatient clinics identified patients who met trial criteria and obtained verbal consent to be approached by the research team. Research personnel either approached the potential participant in the clinic or entered electronic patient records to obtain their contact information. Informed consent was obtained in person or virtually.

This trial was advertised to CHF and CKD patients on patient education websites, on posters in participating outpatient clinics, and through mass emails. Patients who contacted the research team through advertising were sent our Referral Form via email to be completed and returned via email by their physician. The Referral Form screened potential participants based on the inclusion and exclusion criteria. Potential participants who qualified for the trial were then directed through the consenting process virtually.

DATA STORAGE

All data is stored on secure servers within the UHN digital environment and will remain there for at least 10 years after study completion.

PRIVACY AND CONFIDENTIALITY

Subjects are issued a tracking number when information regarding any identifying information is transmitted for analysis. Subject anonymity and confidentiality is preserved. Only aggregate data will be published.

All research personnel have signed an employee confidentiality agreement ensuring that confidential information is not disclosed to any other person or entity. All source documents containing personal identifiers are stored in filing cabinets under lock and key. The database is stored electronically on the firewall-protected server, making it inaccessible externally. Access to the room, which contains the research file server, is restricted to designated persons who are employed by the Cardiac eHealth laboratory at the UHN.

Discussion of the study with persons outside the research team will never reveal personal identifiers of participants. All access to data is denied to persons outside the research team. Data transmission will occur via encrypted storage material over the Internet.

ELIGIBILITY:
Inclusion criteria:

* Biological males and females who are 18 years
* Diagnosed with CHF, including reduced (≤ 40%), mid-range (≥ 41 and ≤ 49%), or preserved (≥ 50%) ejection fraction based on New York Heart Association Classes 2 to 4 (NYHA II-IV) for 3 or more months prior to enrollment, OR diagnosed with advanced CKD (> 10% risk of requiring dialysis within 2 years using the 4-variable, 2-year Kidney Failure Risk equation) or end-stage renal disease and on dialysis
* Oral and written comprehension of English
* Personal access to an email address, a computer, and the Internet
* Informed written consent

Exclusion criteria:

* Scheduled for advanced surgical therapy (e.g., transplantation) within 3 months of enrollment
* Record of significant comorbidities at enrollment that is expected to prohibit full participation (e.g., dementia, psychosis, or severe depression)
* Life expectancy < 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (18 years or older) biologically-born males and females diagnosed with CHF or CKD and fluent in English, with access to a computer, email address, and the Internet
Sampling Method: Non-Probability Sample
Enrollment: 215 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2023-01-16 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Self-reported overall mental health | Baseline and study completion (up to 16 months)
  The primary goal of the study is to evaluate whether engagement with ODYSSEE-vCHAT significantly changes from baseline the proportion of participants with clinically improved or sustained positive mental health (defined as a "minimally important increase" of at least 3.8 points or a score of at least 65 on the MCS) at study completion.

SECONDARY OUTCOMES:
Self-reported depression | Baseline, months 4 and 8, and study completion (up to 16 months)
  9-Item Patient Health Questionnaire (PHQ-9)
Self-reported anxiety | Baseline, months 4 and 8, and study completion (up to 16 months)
  7-Item Generalized Anxiety Disorder (GAD-7)
Self-reported loneliness | Baseline, months 4 and 8, and study completion (up to 16 months)
  6-Item Revised UCLA Loneliness Scale (RULS-6)
Self-reported psychological wellbeing | Baseline, months 4 and 8, and study completion (up to 16 months)
  Flourishing Scale (FS)
Self-reported CHF health-related quality of life | Baseline, months 4 and 8, and study completion (up to 16 months)
  12-Item Kansas City Cardiomyopathy Questionnaire (KCCQ-12)
Self-reported CKD health-related quality of life | Baseline, months 4 and 8, and study completion (up to 16 months)
  36-Item Kidney Disease Quality of Life Instrument (KDQOL-36)
Self-reported engagement in goal-directed activities for living well | Baseline, months 4 and 8, and study completion (up to 16 months)
  Evaluation of Goal-Directed Behaviours to Promote Well-Being and Health (EUROIA), developed by the principal investigator
Self-reported adherence to self-care behaviours (CHF only) | Baseline, months 4 and 8, and study completion (up to 16 months)
  9-Item European Heart Failure Self-care Behaviour scale (EHFScB-9)
Self-reported active involvement in medical care | Baseline, months 4 and 8, and study completion (up to 16 months)
  6-Item Self-Efficacy for Managing Chronic Disease (SEMCD-6)
Self-reported social support | Baseline, months 4 and 8, and study completion (up to 16 months)
  ENRICHD Social Support Instrument (ESSI)
Self-reported physical functioning | Baseline, months 4 and 8, and study completion (up to 16 months)
  Godin-Shepard Leisure-Time Physical Activity Questionnaire (GSLTPAQ)
Self-reported alcohol, nicotine, and cannabis use | Baseline, months 4 and 8, and study completion (up to 16 months)
  Alcohol, Smoking and Substance Involvement Screening Test (ASSIST)
Engagement with self-care resources | Baseline, months 4 and 8, and study completion (up to 16 months)
  Sum login minutes, sum logins, and number of login days prior to a login lapse ≥ 1 month

OTHER OUTCOMES:
Gender interactions | Baseline, months 4 and 8, and study completion (up to 16 months)
  Exploratory analyses will be conducted for gender categories represented by participants (male, female, gender fluid or non-binary, and not specified).

CONTACTS AND LOCATIONS:
Overall Officials: Robert P Nolan, PhD, Principal Investigator — University Health Network, Toronto
Locations (4):
- Canada (4):
  - The Ottawa Hospital, Ottawa, Ontario
  - University Health Network, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rutledge T, Reis VA, Linke SE, Greenberg BH, Mills PJ. Depression in heart failure a meta-analytic review of prevalence, intervention effects, and associations with clinical outcomes. J Am Coll Cardiol. 2006 Oct 17;48(8):1527-37. doi: 10.1016/j.jacc.2006.06.055. Epub 2006 Sep 26. PMID 17045884
- [Background] Celano CM, Villegas AC, Albanese AM, Gaggin HK, Huffman JC. Depression and Anxiety in Heart Failure: A Review. Harv Rev Psychiatry. 2018 Jul/Aug;26(4):175-184. doi: 10.1097/HRP.0000000000000162. PMID 29975336
- [Background] Watnick S, Wang PL, Demadura T, Ganzini L. Validation of 2 depression screening tools in dialysis patients. Am J Kidney Dis. 2005 Nov;46(5):919-24. doi: 10.1053/j.ajkd.2005.08.006. PMID 16253733
- [Background] Murtagh FE, Addington-Hall J, Higginson IJ. The prevalence of symptoms in end-stage renal disease: a systematic review. Adv Chronic Kidney Dis. 2007 Jan;14(1):82-99. doi: 10.1053/j.ackd.2006.10.001. PMID 17200048
- [Background] Hoang VL, Green T, Bonner A. Informal caregivers' experiences of caring for people receiving dialysis: A mixed-methods systematic review. J Ren Care. 2018 Jun;44(2):82-95. doi: 10.1111/jorc.12235. Epub 2018 Jan 22. PMID 29357407
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Ware P, Ross HJ, Cafazzo JA, Boodoo C, Munnery M, Seto E. Outcomes of a Heart Failure Telemonitoring Program Implemented as the Standard of Care in an Outpatient Heart Function Clinic: Pretest-Posttest Pragmatic Study. J Med Internet Res. 2020 Feb 8;22(2):e16538. doi: 10.2196/16538. PMID 32027309
- [Background] Lakkireddy DR, Chung MK, Gopinathannair R, Patton KK, Gluckman TJ, Turagam M, Cheung JW, Patel P, Sotomonte J, Lampert R, Han JK, Rajagopalan B, Eckhardt L, Joglar J, Sandau KE, Olshansky B, Wan E, Noseworthy PA, Leal M, Kaufman E, Gutierrez A, Marine JE, Wang PJ, Russo AM. Guidance for cardiac electrophysiology during the COVID-19 pandemic from the Heart Rhythm Society COVID-19 Task Force; Electrophysiology Section of the American College of Cardiology; and the Electrocardiography and Arrhythmias Committee of the Council on Clinical Cardiology, American Heart Association. Heart Rhythm. 2020 Sep;17(9):e233-e241. doi: 10.1016/j.hrthm.2020.03.028. Epub 2020 Apr 1. PMID 32247013
- [Background] Manemann SM, Chamberlain AM, Roger VL, Griffin JM, Boyd CM, Cudjoe TKM, Jensen D, Weston SA, Fabbri M, Jiang R, Finney Rutten LJ. Perceived Social Isolation and Outcomes in Patients With Heart Failure. J Am Heart Assoc. 2018 May 23;7(11):e008069. doi: 10.1161/JAHA.117.008069. PMID 29794038
- [Background] Moorthi RN, Latham-Mintus K. Social isolation in chronic kidney disease and the role of mobility limitation. Clin Kidney J. 2019 Jan 14;12(4):602-610. doi: 10.1093/ckj/sfy134. eCollection 2019 Aug. PMID 31384455
- [Background] Bajwah S, Wilcock A, Towers R, Costantini M, Bausewein C, Simon ST, Bendstrup E, Prentice W, Johnson MJ, Currow DC, Kreuter M, Wells AU, Birring SS, Edmonds P, Higginson IJ. Managing the supportive care needs of those affected by COVID-19. Eur Respir J. 2020 Apr 23;55(4):2000815. doi: 10.1183/13993003.00815-2020. Print 2020 Apr. PMID 32269090
- [Background] Reza N, DeFilippis EM, Jessup M. Secondary Impact of the COVID-19 Pandemic on Patients With Heart Failure. Circ Heart Fail. 2020 May;13(5):e007219. doi: 10.1161/CIRCHEARTFAILURE.120.007219. Epub 2020 Apr 30. No abstract available. PMID 32352841
- [Background] Rolland B, Haesebaert F, Zante E, Benyamina A, Haesebaert J, Franck N. Global Changes and Factors of Increase in Caloric/Salty Food Intake, Screen Use, and Substance Use During the Early COVID-19 Containment Phase in the General Population in France: Survey Study. JMIR Public Health Surveill. 2020 Sep 18;6(3):e19630. doi: 10.2196/19630. PMID 32589149
- [Background] Juniper EF, Guyatt GH, Willan A, Griffith LE. Determining a minimal important change in a disease-specific Quality of Life Questionnaire. J Clin Epidemiol. 1994 Jan;47(1):81-7. doi: 10.1016/0895-4356(94)90036-1. PMID 8283197
- [Background] Ware JE Jr. SF-36 health survey update. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3130-9. doi: 10.1097/00007632-200012150-00008. No abstract available. PMID 11124729
- [Background] Chung ML, Moser DK, Lennie TA, Frazier SK. Perceived social support predicted quality of life in patients with heart failure, but the effect is mediated by depressive symptoms. Qual Life Res. 2013 Sep;22(7):1555-63. doi: 10.1007/s11136-012-0294-4. Epub 2012 Oct 18. PMID 23076798
- [Background] Sakakibara BM, Ross E, Arthur G, Brown-Ganzert L, Petrin S, Sedlak T, Lear SA. Using Mobile-Health to Connect Women with Cardiovascular Disease and Improve Self-Management. Telemed J E Health. 2017 Mar;23(3):233-239. doi: 10.1089/tmj.2016.0133. Epub 2016 Sep 13. PMID 27623231
- [Background] van Woudenberg TJ, Simoski B, Fernandes de Mello Araujo E, Bevelander KE, Burk WJ, Smit CR, Buijs L, Klein M, Buijzen M. Identifying Influence Agents That Promote Physical Activity Through the Simulation of Social Network Interventions: Agent-Based Modeling Study. J Med Internet Res. 2019 Aug 5;21(8):e12914. doi: 10.2196/12914. PMID 31381504
- [Background] Beishuizen CR, Stephan BC, van Gool WA, Brayne C, Peters RJ, Andrieu S, Kivipelto M, Soininen H, Busschers WB, Moll van Charante EP, Richard E. Web-Based Interventions Targeting Cardiovascular Risk Factors in Middle-Aged and Older People: A Systematic Review and Meta-Analysis. J Med Internet Res. 2016 Mar 11;18(3):e55. doi: 10.2196/jmir.5218. PMID 26968879
- [Background] Nolan RP, Ross HJ, Farkouh ME, Huszti E, Chan S, Toma M, D'Antono B, White M, Thomas S, Barr SI, Perreault S, McDonald M, Zieroth S, Isaac D, Wielgosz A, Mielniczuk LM. Automated E-Counseling for Chronic Heart Failure: CHF-CePPORT Trial. Circ Heart Fail. 2021 Jan;14(1):e007073. doi: 10.1161/CIRCHEARTFAILURE.120.007073. Epub 2021 Jan 19. PMID 33464959
- [Background] Kroenke K, Spitzer RL, Williams JB, Lowe B. The Patient Health Questionnaire Somatic, Anxiety, and Depressive Symptom Scales: a systematic review. Gen Hosp Psychiatry. 2010 Jul-Aug;32(4):345-59. doi: 10.1016/j.genhosppsych.2010.03.006. Epub 2010 May 7. PMID 20633738
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Wongpakaran N, Wongpakaran T, Pinyopornpanish M, Simcharoen S, Suradom C, Varnado P, Kuntawong P. Development and validation of a 6-item Revised UCLA Loneliness Scale (RULS-6) using Rasch analysis. Br J Health Psychol. 2020 May;25(2):233-256. doi: 10.1111/bjhp.12404. Epub 2020 Jan 30. PMID 31999891
- [Background] Vaglio J Jr, Conard M, Poston WS, O'Keefe J, Haddock CK, House J, Spertus JA. Testing the performance of the ENRICHD Social Support Instrument in cardiac patients. Health Qual Life Outcomes. 2004 May 13;2:24. doi: 10.1186/1477-7525-2-24. PMID 15142277
- [Background] Lorig KR, Sobel DS, Ritter PL, Laurent D, Hobbs M. Effect of a self-management program on patients with chronic disease. Eff Clin Pract. 2001 Nov-Dec;4(6):256-62. PMID 11769298
- [Background] Hays RD, Kallich JD, Mapes DL, Coons SJ, Carter WB. Development of the kidney disease quality of life (KDQOL) instrument. Qual Life Res. 1994 Oct;3(5):329-38. doi: 10.1007/BF00451725. PMID 7841967
- [Background] Green CP, Porter CB, Bresnahan DR, Spertus JA. Development and evaluation of the Kansas City Cardiomyopathy Questionnaire: a new health status measure for heart failure. J Am Coll Cardiol. 2000 Apr;35(5):1245-55. doi: 10.1016/s0735-1097(00)00531-3. PMID 10758967
- [Background] Kaczorowski J, Chambers LW, Dolovich L, Paterson JM, Karwalajtys T, Gierman T, Farrell B, McDonough B, Thabane L, Tu K, Zagorski B, Goeree R, Levitt CA, Hogg W, Laryea S, Carter MA, Cross D, Sabaldt RJ. Improving cardiovascular health at population level: 39 community cluster randomised trial of Cardiovascular Health Awareness Program (CHAP). BMJ. 2011 Feb 7;342:d442. doi: 10.1136/bmj.d442. PMID 21300712
- [Background] Amireault S, Godin G, Lacombe J, Sabiston CM. The use of the Godin-Shephard Leisure-Time Physical Activity Questionnaire in oncology research: a systematic review. BMC Med Res Methodol. 2015 Aug 12;15:60. doi: 10.1186/s12874-015-0045-7. PMID 26264621
- [Background] Diener E, Wirtz D, Tov W, Kim-Prieto C, Choi D, Oishi S, Biswas-Diener R. New measures of well-being: Flourishing and positive and negative feelings. Social Indicators Research. 2009; 39: 247-66.
- [Background] Jaarsma T, Arestedt KF, Martensson J, Dracup K, Stromberg A. The European Heart Failure Self-care Behaviour scale revised into a nine-item scale (EHFScB-9): a reliable and valid international instrument. Eur J Heart Fail. 2009 Jan;11(1):99-105. doi: 10.1093/eurjhf/hfn007. PMID 19147463
- See also: COVID-19 fears may be responsible for a 'dramatic drop' in cardiac patients seeking care. — https://www.ctvnews.ca/health/covid-19-fears-possible-reason-for-dramatic-drop-in-cardiac-patients-seeking-care-doctors-1.4897720